CLINICAL TRIAL: NCT00468429
Title: Comparative Study of the Safety and Effectiveness Between Off-Label Subconjunctival Bevacizumab and Mitomycin C in Glaucoma Filtering Surgery.
Brief Title: Subconjunctival Bevacizumab to Prevent Bleb Failure After Glaucoma Filtration Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grewal Eye Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEI-00001
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; Bevacizumab; Glaucoma Filtration Surgery; Mitomycin C; Intraocular Pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Subconjunctival Bevacizumab

SUMMARY:
This study analyzes the safety and efficacy of off-label Subconjunctival Injection of bevacizumab (Avastin) versus 0.02% mitomycin C (MMC) for preventing bleb failure following glaucoma filtration surgery.

DETAILED DESCRIPTION:
Glaucoma Filtration Surgery (GFS) remains the definitive surgical management for elevated IOL uncontrolled by medical management. Bleb failure is a major factor limiting the longterm success of trabeculectomy surgery. Bleb failure involves vascularization with fibroblast migration and eventual scarring of the fistula tract. Vascular Endothelial Growth Factor (VEGF) is a unique mitogen specific to vascular endothelial cells and the signal cascade leading to fibroblast migration and proliferation involves dynamic interaction between many proteins. Blocking the neovascular signal cascade with anti-VEGF molecules like Bevacizumab may lead to a decrease in fibroblast proliferation by decreasing the supply of mitogenic cytokines such as fibroblast growth factor (FGF) carried in by new vessel formation and decreasing the known synergism that exists between VEGF and fibroblast growth factor (FGF) The study is designed as an off-label, randomized, parallel, comparative study. Patients who meet the inclusion/exclusion criteria and sign the informed consent will be included. After enrollment, patients will be randomized into two groups: trabeculectomy with off-label subconjunctival bevacizumab or trabeculectomy with mitomycin-C.This study aims to compare the safety and effectiveness of off-label subconjunctival bevacizumab and subtenon Mitomycin C in glaucoma filtration surgery (GFS). The primary endpoint is to prove the effectiveness via the reduction of IOP and grading of bleb photographs according to the Moorfields Bleb Grading Protocol, and the secondary endpoint is to prove the safety via the incidence of complications and adverse events.

Procedure: Surgical technique Trabeculectomy will be performed after the administration of retrobulbar or peribulbar anesthesia with lidocaine. For the limbus-based procedure, a bridle suture (4-0 silk) will be placed under the superior rectus muscle tendon, and the conjunctiva and Tenon's capsule will be incised in the superior quadrant 8 to 10 mm posterior to the surgical limbus. The conjunctiva and Tenon's capsule will be dissected anterior to the limbus. Meticulous hemostasis will be achieved with bipolar cautery. In cases randomized to MMC usage, a cellulose sponge (approximately 6 × 12 mm × 1 mm) soaked with mitomycin C (0.2 mg/ml) will be applied over the intended site of the scleral flap for 1 to 3 minutes. The duration of mitomycin C application will be based on the preoperative evaluation of each patient's risk factors for failure. Copious irrigation with balanced salt solution will be performed to wash away residual MMC. A ½ to 2/3 thickness square scleral flap (approximately 3.5 × 3.5 mm) will be then dissected into the clear cornea. After resection of an anterior trabecular block (approximately 2.5 × 1 mm), an iridectomy will be performed. The scleral flap will be sutured with two or three 10-0 nylon sutures at its corners. The conjunctiva and Tenon's capsule will be closed in a single continuous layer with 8-0 Vicryl suture. In the subjects randomized to receive Injection Bevacizumab, 0.05 ml of reconstituted bevacizumab drug (1.25 mg) will be injected subconjunctivally adjacent to the bleb. Atropine eye ointment will be placed in the fornix and the eye will be patched. In the early postoperative period, all patients will be treated with topical corticosteroids (four times daily) for two weeks, which will be tapered-off slowly over six to eight weeks. Suture-lysis with argon laser will be performed under topical anesthesia when, in the opinion of the surgeon, filtration is judged to be too low and the IOP too high for the patient to meet the target pressure.

Preparation of the Drug:

Bevacizumab Avastin (Avastin) is available in a sterile vial (100 mg in 4 ml) preservative free and in order to ensure safety the vial injection will be administered within one day.

Subconjunctival Injections (1.25mg drug in 0.05ml) will be given at the end of the surgery adjacent to the bleb raised using a single-use 30-gauge needle and a tuberculin syringe.

Follow-Up: The following demographic and clinical data will be extracted from the medical records of eligible patients: race, age of the patient at the time of surgery, gender, eye laterality, preoperative visual acuity, refractive error, average of IOP readings during three months before surgery, number of medications recorded during the three months preceding trabeculectomy, concurrent ocular diseases before or at the time of surgery, history of intraocular or extraocular surgery that involved the conjunctiva, previous laser surgery for glaucoma (argon laser trabeculoplasty, iridoplasty, or peripheral iridotomy), visual field mean deviation of the last field before surgery, date of surgery, type of conjunctival flap, concentration and duration of mitomycin C application, site and dose of subconjunctival Bevacizumab injection and intraoperative complications.

Postoperative IOP, number of medications, visual acuity, complications, postoperative suture lysis, and surgery performed after trabeculectomy will be recorded. At each visit, the examination will include measurement of Snellen best corrected visual acuity (BCVA), IOP using a calibrated applanation tonometer, slit-lamp biomicroscopy, Seidel testing, and ophthalmoscopy. Humphrey perimetry (24-2 or 10-2) will be done prior to surgery, at 3 and 6 months post intervention to assess for objective disease progression. There will be 7 post-operative and follow-up visits within 6 months of surgery: postoperative days 1, 7, 14, 30, 60, 90 and 180. A window of ± 7 days is allowed for the 30, 60, 90 day visits and ± 14 days for the 180 day visits. On each visit Bleb photographs would be recorded and graded according to the Moorfields Bleb Grading Protocol by a single observer.

Outcomes:

Complete success will be defined as an IOP < 18mmHg without anti- glaucoma medications at 6 months follow up after surgery or at least a 20% reduction from baseline IOP.

Qualified Success will be defined as an IOP of <18mmHg with one anti-glaucoma medication.

Failure will be defined as IOP >21 mmHg or not reduced by 20% below baseline on two consecutive follow-up visits after three months despite medication, IOP ≤5 mmHg on two consecutive follow-up visits after three months, additional glaucoma surgery, or loss of light perception.

Eyes that will be Seidel positive within the first month of follow-up will be classified as wound leaks, and those occurring after one month will be categorized as bleb leaks. Cataracts will be considered to have progressed if there is loss of ≥2 lines of Snellen BCVA that is attributed to the cataract at the six-month follow-up visit or after, or if cataract surgery is performed.

Statistical analysis Univariate comparisons between treatment groups will be made by the two-sided Student t test, χ2 test, or Fisher exact test. The association of surgical complications with treatment outcome, vision loss, and cataract progression will be assessed for statistical significance with the χ2 test or Fisher exact test. A p value of .05 or less will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years or over.
2. Patient with uncontrolled intraocular pressure on maximum tolerated medical therapy (both primary open angle and primary angle closure glaucoma), requiring trabeculectomy.
3. Indications for surgery are based on our own practice patterns: (1) IOP values that are associated with high probability of glaucoma progression and (2) deterioration of the visual field or changes of the optic disk that is compatible with progressive glaucomatous damage, as judged by the examining physician.
4. No history of prior surgical procedure like trabeculectomy, cataract surgery, posterior segment surgery etc.
5. Subject able and willing to cooperate with investigation plan.
6. Subject able and willing to complete postoperative follow-up requirements.
7. Subject willing to sign informed consent form.

Exclusion Criteria:

1. Known allergic reaction to mitomycin-C/ bevacizumab.
2. Subject is on warfarin and discontinuation is not recommended.
3. Normal tension glaucoma.
4. Participation in an investigational study during the 30 days preceding trabeculectomy
5. Patients who had undergone major surgery utpo 28 days before.
6. Ocular infection within 14 days prior to trabeculectomy.
7. Pregnant or breast-feeding women.
8. Patients with uncontrolled diabetes and hypertension or any other medical condition that increase the risk of complications

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
IOP < 18mmHg without anti- glaucoma medications at 6 months follow up after surgery or at least a 20% reduction from baseline IOP. | 6 months

SECONDARY OUTCOMES:
adverse reaction to bevacizumab at site of injection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Jain, MD, Principal Investigator — Grewal Eye Institute; SPS Grewal, MD, Study Chair — Grewal Eye Institute; Gagandeep S Brar, MD, Study Director — Grewal Eye Institute; Dilraj S Grewal, MBBS, Study Director — Grewal Eye Institute
Locations (1):
- Grewal Eye Institute, Chandigarh, Chandigarh, India